CLINICAL TRIAL: NCT05461586
Title: Clinical Investigation of Refraction Techniques
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MDEV104MREE
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MR #1/MR #2: Subjects who participated in PCOL-102-AHSF who were bilaterally implanted with TECNIS IOL lenses will be randomized into the (MR #1/MR #2) sequence and receive two different maximum refractive techniques one at a time consecutively.
  Interventions: Device: Refractive Technique (MR #1); Device: Refractive Technique (MR #2)
- MR#2/MR#1: Subjects who participated in PCOL-102-AHSF who were bilaterally implanted with TECNIS IOL lenses will be randomized into the (MR#2/MR#1) sequence and receive two different maximum refractive techniques one at a time consecutively.
  Interventions: Device: Refractive Technique (MR #1); Device: Refractive Technique (MR #2)

INTERVENTIONS:
Device: Refractive Technique (MR #1) — Fogging method that employs fogging lens to ensure there is sufficient visual defocus to induce blur.
Device: Refractive Technique (MR #2) — Duochrome method that employs the chromatic aberration of the eye, with the shorter wavelengths (green) focused in front of the longer (red) wavelengths

SUMMARY:
Prospective, multi-center, non-interventional, randomized, comparative clinical study to identify an optimal refractive technique that provides maximum plus refractive endpoint for best corrected distance visual acuity (BCDVA).

ELIGIBILITY:
Inclusion Criteria:

1. Participant in PCOL-102-AHSF who were bilaterally implanted with TECNIS IOL, Models C1V000, C2V000 or ICB00 and have completed and are at least 30 days postoperative from their second eye surgery;
2. At least one implanted eye with clear ocular media;
3. Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in Australia and New Zealand;
4. Availability, willingness and sufficient cognitive awareness to comply with examination procedures.

Exclusion Criteria:

1. Best-corrected distance visual acuity (BCDVA) worse than 0.66 decimal (6/9 or 20/30 Snellen);
2. Subjects with ongoing adverse events that might impact outcomes during the study visit as determined by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participant in PCOL-102-AHSF who were bilaterally implanted with TECNIS IOL, Models C1V000, C2V000 or ICB00 and have completed and are at least 30 days postoperative from their second eye surgery.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Difference between two manifest refractive techniques on outcome variable MRSE | Day 0
  Refractive technique 1 will use a plus lens fogging technique and refractive technique 2 will use the Duochrome technique to achieve maximum plus refraction for best-corrected visual acuity (BCDVA).
Difference between two manifest refractive techniques on visual acuity | Day 0
  Refractive technique 1 will use a plus lens fogging technique and refractive technique 2 will use the Duochrome technique to achieve maximum plus refraction for best-corrected visual acuity (BCDVA).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (1):
- Sunshine Eye Clinic, Birtinya, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu